CLINICAL TRIAL: NCT05280613
Title: The Family Check-Up: Implementing a New Family-Centred Model Within Autism Services
Brief Title: The Family Check-Up in Autism Services
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Teresa Bennett, Child and Adolescent Psychiatrist; Associate Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FAIR Study
Record Dates: First submitted 2021-12-21; First posted 2022-03-15 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Autism Spectrum Disorder; Behavior Problem; Emotional Problem
MeSH Terms: conditions — Autism Spectrum Disorder; Mental Disorders | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: An intention-to-treat, parallel-arm randomized controlled trial of N=80 autistic children/youth (ages 6-17 years) with ASD and high levels of EBP and their caregivers.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants will know whether they have been randomized to receive the Family Check-Up or treatment as usual. Clinicians cannot be blinded because they will be providing the intervention. However, investigators and outcome assessors will be blinded to treatment status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Family Check-Up (Experimental): Families randomized to the Family Check-Up arm will be connected with a clinician who will provide the Family Check-Up. The Family Check-Up® (FCU) is an ecologically sensitive, evidence-based intervention that was developed to decrease childhood EBP by 1) assessing known ecological (child, family and contextual) risk and protective factors; 2) engaging parents in a tailored plan to enhance positive parenting and family management skills; and 3) connecting families to a tailored suite of child and family services and supports. Services may include an evidence-based suite of parenting sessions ("Everyday Parenting Curriculum [EPC]") created by FCU developers for direct tailoring to the FCU feedback session.
  Interventions: Behavioral: Family Check-Up
- Treatment as Usual (Active Comparator): Treatment as Usual participants will be connected to a Family Service Coordinator within the Autism Program, who can direct the family to appropriate services and resources. Services may include consultation on child behaviours, workshops on various topics, parenting programs, Applied Behaviour Analysis, support groups, and group recreational programs. Families in the treatment as usual arm will be offered the Family Check-Up upon completion of the study.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Family Check-Up — See arm/group description
  Arms: Family Check-Up
Behavioral: Treatment as Usual — See arm/group description
  Arms: Treatment as Usual

SUMMARY:
Many children and youth with autism spectrum disorder have high levels of emotional and behavioural problems. Parents play a powerful role in supporting their children's well-being. Research also shows that certain factors (e.g., parent mental health, access to services) can affect autistic children's well-being in important ways. Despite this, autism services rarely ask about, or act upon, the factors that we know affect child and family well-being. We are addressing this problem by testing a program called the Family Check-Up within a large autism service. The Family Check-Up is a strengths-based, family-centred program aimed at improving child well-being by working with parents to identify their family's unique strengths and challenges, set goals for change, strengthen positive parenting, and connect to needed supports.

DETAILED DESCRIPTION:
Prevalence rates of emotional and behavior problems (EBP) in children and youth with autism spectrum disorder (ASD) are high (40-70%), and often cause severe and chronic impairment. Childhood EBP has been linked to ecological adversity (e.g., social isolation, parenting stress). Positive parenting practice can protect against adverse child outcomes such as poor self-regulation, chronic stress and EBP. Interventions aspiring to alleviate EBP in children with ASD need to involve caregivers in a collaborative, empowering and meaningful way.

In the current Ontario ASD services landscape, there are no evidence-based family-centered programs that adequately address these needs. The Family Check-Up (FCU) is a brief, ecologically sensitive, evidence-based, trans-diagnostic intervention that engages families in a process of enhancing positive parenting practices to reduce child EBP. It is unique in its multi-modal assessment of ecological risk and protective factors, strength-based motivational interviewing approach and health maintenance design, providing annual check-ups during key periods of development. It may be linked to an optional, tailored "Everyday Parenting Curriculum" (EPC). Studies have demonstrated sustained, reliable, and robust positive effects on child EBP, caregiver depression, and positive parenting practices in other populations at risk, but the FCU has not been evaluated in families of autistic children and youth. Thus, the objective is to evaluate FCU implementation in the Hamilton Health Sciences (HHS) Autism Program, with delivery by autism therapists, in order to demonstrate sustainable effectiveness within real-world settings.

ELIGIBILITY:
Inclusion Criteria:

* Child 6-17 years of age with a confirmed diagnosis of ASD
* Enrollment in the Ontario Autism Program
* Minimum developmental age of 2
* Elevated emotional and behaviour problems
* Residing with the same caregiver at least 5 days/week or every other week for the past 2 months and foreseeable future

Exclusion Criteria:

* Parent with insufficient knowledge of English to complete assessments
* Current enrollment in another intervention study
* Active significant safeguarding concerns (e.g., child acute severe self-harm or aggression, acute parent or child suicidality)
* Prior participation in the Family Check-Up

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2025-02-11 (Actual)

PRIMARY OUTCOMES:
Change in Aberrant Behavior Checklist (ABC) - irritability subscale | 0, 3, 6 months
  The ABC was designed to measure psychiatric symptoms and behavioural disturbances. The irritability subscale is commonly used as an outcome in ASD research. Scores can range from 0 - 45, with higher scores indicating higher irritability
Change in Home Situation Questionnaire -ASD (HSQ-ASD) | 0, 3, 6 months
  The HSQ-ASD was designed to measure the severity of non-compliant behaviour of autistic children in common situations

SECONDARY OUTCOMES:
Change in Center for Epidemiological Studies Depression Scale - Revised (CESD-R) | 0, 3, 6 months
  The CESD-R is a 20 item measure of depression. Scores range from 0-80 with higher scores indicating worse depression.
Change in Generalized Anxiety Disorder-7 (GAD-7) | 0, 3, 6 months
  The GAD-7 is a brief measure of generalized anxiety. Scores range from 0-21 with higher scores indicating greater anxiety
Change in Parenting Daily Hassles | 0, 3, 6 months
  The Parenting Daily Hassles is a measure of parenting stress. Scores range from 0 - 80 with higher scores indicating greater parenting stress.
Change in Parenting Young Children (PARYC) | 0, 6 months
  This is a measure of important parenting skills such as positive behaviour support, limit setting, and proactive parenting. Scores range from 0 - 72, with higher scores indicating higher use of parenting skills
Change in Parental Monitoring Scale | 0, 6 months
  This is a measure of monitoring, an important parenting skill. Scores range from 0-44 with higher scores indicating higher monitoring.
Change in Parent Empowerment and Efficacy Measure (PEEM) | 0, 6 months
  This is a measure of parents' sense of control or capacity to manage the challenges of being a parent and provide a safe and supportive home environment. Scores range from 20-200 and higher scores indicate higher parent empowerment and efficacy.
Change in Brief Coping Orientation to Problems Experienced (Brief COPE) | 0, 6 months
  This is a measure of coping strategies. Scores range from 28 - 112 with higher scores indicating higher usage of coping strategies.
Clinical Global Impressions - Improvement (CGI-I) | 0, 3, 6 months
  The CGI-I measures the change in problem behaviours over time. Scores of 1-3 indicate improvement; a score of 4 indicates no change, and scores of 5-7 indicate worsening of behaviour.

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dishion TJ, Mauricio AM. The Family Check-Up model as prevention and treatment of adolescent drug use: The intervention strategy, outcomes, and implementation model. In: Family-Based Prevention Programs for Children and Adolescents (pp. 98-122). London, UK: Psychology Press: 2015.
- [Background] Dishion TJ, Stormshak EA, Kavanagh KA. Everyday parenting: A professional's guide to building family management skills. Champaign, IL: Research Press; 2012.
- [Background] Aman MG, Singh NN, Stewart AW, Field CJ. Psychometric characteristics of the aberrant behavior checklist. Am J Ment Defic. 1985 Mar;89(5):492-502. PMID 3158201
- [Background] Kaat AJ, Lecavalier L, Aman MG. Validity of the aberrant behavior checklist in children with autism spectrum disorder. J Autism Dev Disord. 2014 May;44(5):1103-16. doi: 10.1007/s10803-013-1970-0. PMID 24165702
- [Background] Kohout FJ, Berkman LF, Evans DA, Cornoni-Huntley J. Two shorter forms of the CES-D (Center for Epidemiological Studies Depression) depression symptoms index. J Aging Health. 1993 May;5(2):179-93. doi: 10.1177/089826439300500202. PMID 10125443
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Crnic KA, Greenberg MT. Minor parenting stresses with young children. Child Dev. 1990 Oct;61(5):1628-37. doi: 10.1111/j.1467-8624.1990.tb02889.x. PMID 2245752
- [Background] McEachern AD, Dishion TJ, Weaver CM, Shaw DS, Wilson MN, Gardner F. Parenting Young Children (PARYC): Validation of a Self-Report Parenting Measure. J Child Fam Stud. 2012 Jun;21(3):498-511. doi: 10.1007/s10826-011-9503-y. PMID 22876108
- [Background] Stattin H, Kerr M. Parental monitoring: a reinterpretation. Child Dev. 2000 Jul-Aug;71(4):1072-85. doi: 10.1111/1467-8624.00210. PMID 11016567
- [Background] Gibaud-Wallston J, Wandersman LP. Parenting Sense of Competence Scale. Mahwah, NJ: Lawrence Erlbaum Associates; 1978.
- [Background] Folkman S, Lazarus RS, Gruen RJ, DeLongis A. Appraisal, coping, health status, and psychological symptoms. J Pers Soc Psychol. 1986 Mar;50(3):571-9. doi: 10.1037//0022-3514.50.3.571. PMID 3701593